CLINICAL TRIAL: NCT06787027
Title: Evaluation of the Effect of Manual Lymphatic Drainage Method on Edema, Pain and Trismus After Impacted Bilateral Mandibular Third Molar Surgery: a Randomized Clinical Trial
Brief Title: Effect of Manual Massage Technique on Swelling, Pain and Mouth Opening After Bilateral Lower Third Molar Surgery
Acronym: wisdom tooth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Onur ŞAHİN, Associate Professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Impacted Third Molar Tooth; Swelling/ Edema; Pain; Trismus
Keywords: impacted lower third molar; 3dMD; Manual Lymphatic Drainage; edema
MeSH Terms: conditions — Edema; Pain; Trismus

STUDY DESIGN:
Intervention Model Description: Split-mouth model
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Lymphatic Drainage technique (Experimental): Following the morning surgery, MLD therapy was administered in the afternoon of the same day by a professional physiotherapist
  Interventions: Procedure: Manual Lymphatic Drainage technique; Procedure: Conventional Treatment group
- Conventional treatment (Experimental): Postoperatively, patients were prescribed antibiotics (amoxicillin with clavulanic acid, 1 g, twice daily), analgesics (paracetamol, 500 mg, twice daily), and mouthwash (chlorhexidine gluconate, three times daily) for five days.
  Interventions: Procedure: Manual Lymphatic Drainage technique; Procedure: Conventional Treatment group

INTERVENTIONS:
Procedure: Manual Lymphatic Drainage technique — Following the morning surgery, manual lymphatic drainage therapy was administered in the afternoon of the same day by a professional physiotherapist.
Procedure: Conventional Treatment group — patients were prescribed antibiotics (amoxicillin with clavulanic acid, 1 g, twice daily), analgesics (paracetamol, 500 mg, twice daily), and mouthwash (chlorhexidine gluconate, three times daily) for five days. Cold application was recommended to all patients.

SUMMARY:
The aim of this study was to evaluate the effect of manual lymphatic drainage on pain, edema and trismus after impacted mandibular third molar surgery.

DETAILED DESCRIPTION:
This study is a randomized controlled split-mouth trial. A total of 46 healthy patients who presented to our department for the extraction of impacted mandibular third molars were included in this study.The inclusion criteria were as follows: presence of pericoronal infection, no recent use of anti-inflammatory medications, symmetrical impactions on both sides, asymptomatic cases, and class 2, position B or C, vertical and mesioangular impactions. Impactions were classified using the Pell and Gregory classification system.

Exclusion criteria included patients who declined participation, pregnant or lactating individuals, patients with penicillin allergies, those with chronic diseases that could affect healing, uncooperative patients. Following the surgery, manual lymphatic drainage therapy was administered in the afternoon of the same day by a professional physiotherapist using the "Vodder" technique. In this study, measurements were conducted by two researchers. Swelling and trismus values were recorded preoperatively (T0), on the 3rd postoperative day (T1), and on the 7th postoperative day (T2). To assess pain, the VAS was used and values were recorded 1, 2, 3 and 7 days postoperatively. In this study, edema was evaluated using the 3dMD FACE SYSTEM (3dMD, Atlanta, GA), which virtually transfers the patient's face into 3D, allowing for the calculation of volume changes.To assess pain, the Visual Analog Scale (VAS) was used.To determine the effect of MLD therapy on postoperative trismus, the distance between the upper and lower incisors was measured using a digital caliper immediately before the operation, as well as on the 3rd and 7th postoperative days

ELIGIBILITY:
Inclusion Criteria:

* good general health conditions;
* presence of bilateral and symmetrical impacted third molars (according to the classifications of Winter and Pell and Gregory);

Exclusion Criteria:

* no clinical evidence of major facial asymmetry;
* use of medication that would influence or alter wound healing;
* temporomandibular joint disorder history;
* smoking

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
postoperative facial swelling | one week
  Facial swelling
  T0-T1 and T0-T2 scans are opened and superimposed through three reference points:
  endocanthion left (inner most point on commissure of left eye fissure), endocanthion right (inner most point on commissure of right eye fissure) and subnasale (mid point of columella).
  After matching, the swelling was calculated by selecting the area of the swelling and subtracting the two images.

SECONDARY OUTCOMES:
Pain | one week
  VAS measure
Mouth opening | one week
  measurement of the maximal distance between the cutting edge of the right maxillary and right mandibular central incisors with a caliper.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Çelebi University, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulu M, Unal N, Sahin O, Kayali Y. Evaluation of the effect of manual lymphatic drainage method on edema, pain and trismus after impacted bilateral mandibular third molar surgery: a randomized clinical trial. BMC Oral Health. 2025 Mar 26;25(1):438. doi: 10.1186/s12903-025-05817-6. PMID 40140780